CLINICAL TRIAL: NCT03331276
Title: Growth and Safety Study of an Infant Formula for Healthy Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Building Block Nutritionals, LLC (Industry)
Collaborators: Paidion Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BBN-IF-001
Record Dates: First submitted 2017-09-21; First posted 2017-11-06 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Infant Development
MeSH Terms: interventions — lepirudin

STUDY DESIGN:
Intervention Model Description: Formula feed infants will be randomized to receive either a new infant formula formulated for healthy term infants (BBN) or a commercially available infant formula for healthy term infants (Brand). Infants will consume the formula for a total of 16-weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a randomized, controlled, double-blind, study of healthy term formula fed (FF) infants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BBN (Experimental): An experimental Infant Formula, Milk-Based Powder with Iron, for healthy term infants 0 to 12 months of age with high Sn-2 Palmitate, Alpha Lactalbumin and Osteopontin to better mimic human milk.
  Interventions: Other: BBN
- Brand (Active Comparator): A Commercially available Infant Formula, for healthy term infants 0 to 12 months of age (Enfamil TM, Milk-Based Powder with Iron)
  Interventions: Other: Brand

INTERVENTIONS:
Other: BBN — BBN to be feed as the sole source of nutrition for 16 weeks to healthy term infants for 16 weeks.
  Other Names: BBN-001
  Arms: BBN
Other: Brand — Brand to be feed as the sole source of nutrition for 16 weeks to healthy term infants for 16 weeks.
  Other Names: Enfamil
  Arms: Brand

SUMMARY:
A goal of infant formula development is to mimic human milk (HM) both in nutrient composition as well as physiologic outcomes. investigators have developed an infant formula for term infants that more closely resembles the composition of human milk. The purpose of this study is to demonstrate that this formulation meets nutritional requirements and supports age appropriate growth of healthy term infants.

DETAILED DESCRIPTION:
This study is a randomized, controlled, double-blind, study of healthy term formula fed (FF) infants. FF infants will be randomized to receive either a experimental infant formula, formulated for healthy term infants (BBN) or a commercially available infant formula for healthy term infants (Brand). Infants will consume the formula for a total of 16-weeks; infant growth, serum markers for inflammation and tolerance to the formulas will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Infants will be eligible to participate if they meet all of the following conditions. At birth the infant must be:

  1. Healthy, term (early term/no less than 37 weeks, 0 days through late term/no greater than 41 weeks, 6 days), singleton infant
  2. Have a birth weight of ≥ 2500 grams

     At the time of the baseline/enrollment visit, infants must be:
  3. Designated as healthy by a physician
  4. ≤14 days post-natal age (Date of Birth = Day 0)
  5. Weight for age ≥ 5th and ≤ 95th percentile for age according to sex-specific World Health Organization (WHO) growth charts
  6. Length for age ≥ 5th and ≤ 95th percentile for age according to sex-specific World Health Organization (WHO) growth charts
  7. Head circumference for age ≥ 5th and ≤ 95th percentile for age according to sex-specific World Health Organization (WHO) growth charts
  8. Weight for length for age ≥ 5th and ≤ 95th percentile for age according to sex-specific World Health Organization (WHO) growth charts
  9. Exclusively consuming and tolerating a cow's milk infant formula at time of enrollment; only infants whose parent(s) or legal guardian(s) have decided to feed infant formula as the sole soure of nutrition, will be approached for potential study enrollment
  10. Have parent(s) or legal guardian(s) who agree to feed the study formula to the study subject as his/her sole source of nutrition for the duration of the study
  11. Have parent(s) or legal guardian(s) who have read and voluntarily signed an Informed Consent form approved by the Institutional Review Board prior to any participation in the study.

Exclusion Criteria:

Infants will be ineligible if they have any of the following conditions that are judged by a physician to interfere with the infant's normal growth, development, and/or tolerance to an infant formula:

1. Show evidence of anatomic and physiologic defects of the respiratory tract, or other congenital defects (as determined by the clinician);
2. Show evidence of chronic hepatic, gastrointestinal, renal, cardiac, pulmonary, or neurological diseases;
3. Have a maternal history with known adverse effects on the fetus and/or the newborn infant, such as diabetes (gestational diabetes is acceptable if infant's birth weight is < 4300 g), active tuberculosis, perinatal infection, or substance abuse
4. Have a family history of cow's milk protein intolerance/allergy
5. Are an infant from a multiple birth (twin, triplet, etc.) -

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Weight gain | 16 weeks
  g/d

SECONDARY OUTCOMES:
Mean stool consistency | Monthly for 16 weeks
  1= watery, 2= runny / soft, 3= musy / soft, 4= formed soft, 5= hard
Mean fussiness score | Monthly 16 weeks
  0= less fussy than normal, 1= about the same level of fussiness as normal, 2= more fussy than normal
Mean gassiness score | Monthly 16 weeks
  0= no gas, 1= slight amount of gas, 2= moderate amout of gas, 3= excessive amount of gas
Mean interleukin - 6 Concentration | at 16 weeks
  IL - 6 ng/ml
Mean interleukin - 10 Concentration | at 16 weeks
  IL - 10 pg/ml
Mean tumor necrosis factor alpha Concentration | at 16 weeks
  TNF - alpha pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Dunn, MD, Study Director — Paidion Research, Inc.
Locations (6):
- United States (6):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Southeastern Pediatric Associates, Dothan, Alabama
  - Norwich Pediatric Group, Norwich, Connecticut
  - Aventiv Research, Grove City, Ohio
  - HMG Pediatrics at Medical Plaza, Bristol, Tennessee
  - Jackson Clinic, Jackson, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yao M, Lien EL, Capeding MR, Fitzgerald M, Ramanujam K, Yuhas R, Northington R, Lebumfacil J, Wang L, DeRusso PA. Effects of term infant formulas containing high sn-2 palmitate with and without oligofructose on stool composition, stool characteristics, and bifidogenicity. J Pediatr Gastroenterol Nutr. 2014 Oct;59(4):440-8. doi: 10.1097/MPG.0000000000000443. PMID 24840511
- [Derived] Fleming SA, Flunkert S, Kvistgaard AS, McGrath J, Glover DK. New infant formulas for healthy term infants: A randomized, controlled, double-blind, multicenter, non-inferiority design safety study. PLoS One. 2025 Dec 17;20(12):e0336689. doi: 10.1371/journal.pone.0336689. eCollection 2025. PMID 41406156